CLINICAL TRIAL: NCT06563206
Title: Comparison of Tenascin-C Value Rates and Functional Outcomes Between Exergame Therapy and Robotic Therapy in Post-Stroke Patients
Brief Title: Exergame and Robotic Therapy Impact on Tenascin-C and Functional Outcome on Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Lecturer, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0208242322
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Paralysis Arm
Keywords: Robotic Rehabilitation; Video-assisted Rehabilitation; Post-Stroke; Functional Outcome; Tenascin-C
MeSH Terms: conditions — Stroke | interventions — Exergaming; Robotics; Congresses as Topic

STUDY DESIGN:
Intervention Model Description: This study will be conducted using parallel design of three different rehabilitation approach with repeated measurements of outcomes, before and after intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator will be masked from the allocation as well as outcome assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Rehabilitation/Conventional (Active Comparator): The conventional exercise therapy group will be given diathermic, electricity modality, hydrotherapy, and therapeutic exercises in the form of muscle stretching, strengthening exercises, transfer exercises, walking exercises, and hand function exercises for 3 times a week within 6 weeks.
  Interventions: Procedure: Conventional
- Exergame (Experimental): Conventional therapy coupled with virtual reality Exergame exercises on the hands for 3 times a week a time 6 weeks
  Interventions: Procedure: Exergame
- Robotic (Experimental): conventional therapy coupled with robotic therapy exercises on the hands for 3 times a week a time of 6 weeks
  Interventions: Procedure: Robotic

INTERVENTIONS:
Procedure: Exergame — Hand Training assisted with Virtual-Reality
  Arms: Exergame
Procedure: Robotic — Hand Training assisted with Robotic Syrebo
  Arms: Robotic
Procedure: Conventional — Hand Training with Physical Therapist
  Arms: Standard Rehabilitation/Conventional

SUMMARY:
This clinical trial aims to compare the effectiveness of Robotic versus Exergame versus Standard therapy to improve hand function among post-stroke patients. The main questions it aims to answer are:

1, Effectiveness of interventions in functional outcome recovery across time 2. Effectiveness of interventions in affecting Tenascin-C level 3. Clinical outcome difference between all interventions

Participants will be allocated into three groups, either a robotic group, exergame group as the main interventions, and standard rehabilitation group as the active comparator. A serial follow-up will be conducted to assess the selected clinical outcome and differences in outcome

DETAILED DESCRIPTION:
1, Research design This research is an experimental study with a randomized controlled trial research design.

2. Study Setting The research will be carried out among post-stroke patients at two teaching hospitals and one physical rehabilitation center in Makassar

3. Procedure

a. Standard Rehabilitation Comprehensive medical management and rehabilitation of disabilities caused by stroke through the neurorehabilitation approach with the aim of optimizing recovery and or modifying existing remaining symptoms so that stroke people are able to carry out functional activities independently, can adapt to the environment and achieve quality life

b. Exergame Physical exercise of the entire body carried out through active video games that require gross motor skills, visual-spatial coordination, balance, and energy expenditure that are proportional to the intensity of moderate physical activity

c. Robotic Therapy Mirror therapy intervention uses the help of robot exoskeletal to move the sick side. A set of mirror therapy exercises, using Syrebo robotics, using 1 set of Activity Daily Living (ADL) training during therapy, and using a mirror that will reflect a healthy side shadow.

4. Time frame the procedure will be conducted in parallel three times per week for a total of six weeks, with two measurements before and after six weeks of training

5. Outcomes

1. motoric ability of upper extremity using Fugl-Meyer Assessment for Upper Extremities (FMA-UE)
2. Dexterity, coordination and response of finger using the Nine Hole Peg Test (NHPT)
3. Hand motor strength with Handgrip dynamometer
4. Level of Tenascin-C in blood serum before and after

   6. Case definition

a. type of stroke determined by radiology imaging b. phase of stroke (acute, sub-acute or chronic) c. cognitive ability measured using mini-mental state examination (MMSE) d. Spasticity measured by the Modified Ashworth Scale (MAS)

7. Procedure

a. The data collected is primary data obtained in accordance with the inclusion criteria.

b. Samples who are willing to become research subjects will undergo interviews, physical examinations, FMA-UE-Hand Motor Domain, handgrip and NHPT examinations. The interview questionnaire in this study will contain a list of patient identities including name, age, marital status, address, educational history, employment history, history of stroke, cognitive examination (MMSE), and self-reported visual ability.

8. Measurement tools

1. The FMA-UE-Hand Motor Domain scoring system is used to evaluate upper extremity motor function in patients with neurological disorders, such as stroke. The scoring system ranges from 0-14, with higher scores indicating better motor function. The FMA-UE-Hand Motor domain assessment system is broken down into several subscales, namely Mass Flexion and Extension movements, followed by functional movements of grasping (Grasp), including Hook Grasp, Thumb Adduction, Pincer Grasp, Cylinder Grasp, and Spherical Grasp. The assessment will get a score of 0 = None or no movement, 1 = Partial or limited movement, and 2 = Full or perfect movement.
2. The NHPT assessment consists of a square board with 9 pegs. At one end of the board, there is a hole for the peg, and at the other end, there is a shallow round plate for holding the peg. NHPT is performed by having the patient take pegs from a container, one at a time, and place them into the holes in a board, as quickly as possible. The patient must then remove the pegs from the holes, one at a time, and reinsert them into the housing. To practice and register initial scores, the test must be started with the unaffected upper limb. The board should be placed in the centre of the patient's body with the housing holding the pegs oriented toward the hand being tested. Only the hand being evaluated should perform the test. The non-evaluated hand is allowed to grip the edge of the board to provide stability. Patients are scored based on the time required to complete the test activity, recorded in seconds. The stopwatch must start from the moment the participant touches the first peg until the last peg touches the container. This assessment requires a board, of wood or plastic, with 9 holes (10 mm diameter, 15 mm depth), spaced 32 mm or 50 mm apart and a stopwatch.
3. Tenascin-C To perform an ELISA for Tenascin-C, the procedure involves preparing samples and standards according to the kit instructions. The samples and standards are added to wells pre-coated with Tenascin-C-specific antibodies and incubated to facilitate binding. Following incubation, the wells are washed to remove any unbound substances. A detection antibody, conjugated with an enzyme, is then added and incubated. After additional washing, a substrate solution is introduced, causing a color change proportional to the amount of Tenascin-C present. The reaction is stopped with an acid solution, and the optical density is measured using a plate reader. The Tenascin-C concentration in the samples is determined by comparing the optical density readings to a standard curve. Typically, Tenascin-C levels are reported in pg/mL, and the assay range and sensitivity depend on the specific kit used. Accurate interpretation requires comparing the sample values to the standard curve to assess Tenascin-C expression levels, which can provide insights into the biological or pathological state being investigated.

   9. Sample Size

   This clinical trial aims to compare the effectiveness of Robotic Therapy, Exergame Therapy, and Standard Therapy in improving hand function among post-stroke patients. Assuming a standard deviation of 26.75, an expected mean difference of 18.72, and a dropout rate of 30%, the sample size is calculated to be 16 participants per group. This calculation is based on a 95% confidence level (Zα = 1.96) and 80% power (Zβ = 0.84) across the three arms.

   10. Proposed Statistical Analysis

   the data will be analyzed using Analysis of Variance/ ANOVA assuming no difference in baseline characteristic. Next, the relationship between continuous values will be assessed using the Pearson correlation test (normally distributed data) or the Spearman test (data not normally distributed) to determine how big the correlation is between these variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients after ischemic or hemorrhagic stroke
* stable hemodynamics and neurologic state.
* Patients have never undergone treatment with any intervention
* Able to watch television with or without glasses from a distance of 1 meter.
* Patients can understand informed consent to participate in research

Exclusion Criteria:

* Patients with a history of seizures or epilepsy.
* Patients with severe cognitive disorders that can interfere with research objectives (MMSE score <24).
* Patients with field deficits or severe vision disorders.
* The patient is unable to sit upright without help.
* Patients with significant pain in the affected upper limb.
* Patients with significant sensory decreases in the upper limb that are affected
* Patients with other medical conditions (musculoskeletal, neuromuscular, cardio respiration) are uncontrolled and are at risk of disrupting the ability to exercise.

Dropout Criteria

* Patients who were declared dead
* Refusing to continue the training session or less < 50% of all sessions.
* Experiencing hemodynamic and neurological disorders during the training program process.
* Experiencing cybersickness twice in successive training sessions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity (FMA-EU) Score | changes of FMA-UE score from pre-intervention to six weeks after intervention
  a motoric assessment with each score range from 0-2 with a total score range from 0-66. Higher score indicates better and free movement
Nine Hole Peg Test Value | changes of NHPT values from pre-intervention to six weeks after intervention
  an assessment for finger dexterity and coordination where the time of the subject to accomplish task will be recorded. Average healthy adult male completed the NHPT in 19.0 seconds (SD 3.2) with the right hand, and in 20.6 seconds (SD 3.9) with the left hand. For healthy adult women, the NHPT was completed in 17.9 seconds (SD 2.8) and 19.6 seconds (SD 3.4) with the right and left hands, respectively.
Handgrip Dynamometer value | changes of handgrip values from pre-intervention to six weeks after intervention
  The handgrip dynamometer measures hand strength, with a typical range of 0 to 100 kg (0 to 220 lb). For men, normal handgrip strength usually falls between 30-60 kg (66-132 lb), while for women it ranges from 20-40 kg (44-88 lb).
Tenascin-C value | changes of Tenascin-C value from pre-intervention to six weeks after intervention
  The normal range of Tenascin-C levels in healthy individuals typically falls between 50 to 200 ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Rumaisah Hasan, MD, Principal Investigator — Hasanuddin University
Locations (2):
- Indonesia (2):
  - Hasanuddin University, Faculty of Medicine, Makassar, South Sulawesi
  - Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi

IPD SHARING:
Plan to Share IPD: No
No To protect the confidentiality, should the data need to share, any de-identified data will be shared for peer-review